CLINICAL TRIAL: NCT02738684
Title: A Small Sample Exploratory Study to Predict Gefitinib' s Efficacy for Late Stage Lung Adenocarcinoma Patients by Plasma Free Nucleic Acids EGFR Gene Mutation Test
Brief Title: A Study to Predict Gefitinib' s Efficacy for Lung Cancer by Plasma Free Nucleic Acids EGFR Gene Mutation Test
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, XIAOTIANDAI, Department of Respiratory Diseases, Southwest Hospital, China
Other Study IDs: pfnaegmt-023
Record Dates: First submitted 2016-03-22; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Lung Adenocarcinoma
Keywords: lung cancer; adenocarcinoma; EGFR; plasma free nucleic acids
MeSH Terms: conditions — Adenocarcinoma of Lung; Lung Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — predict gefitinib' s efficacy for late stage lung adenocarcinoma patients by plasma free nucleic acids EGFR gene mutation test
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- lung cancer: A small sample exploratory study to predict gefitinib' s efficacy for late stage lung adenocarcinoma patients by plasma free nucleic acids EGFR gene mutation test

SUMMARY:
This project aims to do a small sample exploratory study, to predict EGFR-TKI targeted therapy gefitinib' s efficacy in late stage lung adenocarcinoma patients (phase IIIB or IV), who have negative tissue EGFR gene mutation, positive plasma free nucleic acid EGFR gene.

DETAILED DESCRIPTION:
Results of the study will clarify that if the circulating tumor DNA (ctDNA) EGFR mutation could be used as a screening method for EGFR-TKI targeted therapy for late stage lung cancer patients, as well as a standard for the therapy efficacy. This study can be used as a standard to assess gefitinib' s efficacy after 8 weeks of treatment in IIIB or stage IV lung cancer through tumor tissue negative, ctDNA positive EGFR mutation.

ELIGIBILITY:
Inclusion Criteria:

* Participants in this research must meet the following criteria: histologic diagnosed of lung adenocarcinoma.
* Late stage (stage IIIB or IV) lung adenocarcinoma according to the International Union against cancer (UICC) the latest version of standard cancer TNM staging.
* tumor tissue EGFR mutation negative, and ctDNA EGFR mutation positive correlated with EGFR TKI sensitivity.
* Participants should have signed and dated on the official informed consent.
* Not less than 18 years old.
* At least 1 lesion can be exactly measured.
* Patients whose plasma free nucleic acids EGFR mutation test were positive, and willing to use gefitinib for therapy by their own expense.

Exclusion criteria:

* Patients already received EGFR-TKI treatment previously.
* Patients have pressure on the spinal cord or brain metastases, no symptom, conditions stabled, do not need to use steroid medications for 4 weeks before the start of the study.
* Patients with clinical evidence of any symptoms of severe or uncontrolled hypertension, for example, researchers believe that patients with uncontrolled hypertension and active bleeding will affect the study reliability.
* Patients with uncontrolled nausea or vomiting, chronic gastrointestinal disease, unable to swallow drugs or underwent major bowel resection may affect the full absorption of gefitinib.
* Patients meet any one of the following heart standard: in static State, 3 times ECG check shows average correction QT period (QTc) >470 msec; clinical abnormal symptom of rhythm, conduction, and static ECG, for example completely left beam conduction block, III degrees conduction block, II degrees conduction block, PR period >250 msec, various factors with risks of extended QTc or rhythm disorders, for example, congestive heart failure, low potassium blood syndrome, congenital long QT Syndrome, direct relatives has long QT syndrome or sudden unexplained death in less than 40 years old, drug combination that may prolong the QT interval.
* Patients Have the following history: ILD, drug-induced ILD, radiation Pneumonitis require steroid treatment, clinically active interstitial lung disease.
* Abnormal marrow reservation or organ function.
* Women who are breastfeeding.
* Fertile male or female, who did not taken effective contraceptive measures, women have been pregnant or breast feeding, or positive pregnancy test prior to study (urine or serum).
* Patients don't agree with the study processes, constraints and requirements, and were evaluated by researchers that can't participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in this research must meet the following criteria: histologic diagnosed of lung adenocarcinoma. Late stage (stage IIIB or IV) lung adenocarcinoma according to the International Union against cancer (UICC) the latest version of standard cancer TNM staging.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
RECIST 1.1 Efficacy assessments | 8 weeks
  Categorisation of objective tumour response assessment at each visit will be based on the RECIST 1.1 criteria of response: CR, PR, SD and PD.

CONTACTS AND LOCATIONS:
Overall Officials: DAI X T, doctor, Principal Investigator — Department of Respiratory Diseases, Souty West Hospital

IPD SHARING:
Plan to Share IPD: Yes